CLINICAL TRIAL: NCT00506610
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Flexible Escalating -Dose, Pilot Analgesic Efficacy Study of T-62 in Subjects With Postherpetic Neuralgia
Brief Title: A Study to Determine if an Investigational Pain Medicine Provides Relief of Chronic Pain After a Shingles Outbreak
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K862-06-2001
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Postherpetic Neuralgia
Keywords: Pain; Postherpetic Neuralgia; Neuralgia, Postherpetic; Shingles; Herpes Zoster; Neuropathic Pain
MeSH Terms: conditions — Neuralgia, Postherpetic; Pain; Herpes Zoster; Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: T-62

SUMMARY:
The purpose of this study is to determine whether T-62 is effective in providing relief of pain that can occur after an individual experiences a shingles outbreak, which is an infection in adults caused by the same virus that causes chicken pox.

ELIGIBILITY:
Inclusion Criteria:

* Has a clinical diagnosis of Postherpetic Neuralgia (PHN)
* Experiencing pain for at least 3 months after the healing of shingles rash
* Has at least a weekly average pain intensity of equal to or greater than 4 out of 10
* Females must not be pregnant or breastfeeding and practicing an acceptable method of birth control, or be surgically sterile or post-menopausal
* Will not consume grapefruit or grapefruit juice during the study

Exclusion Criteria:

* Has a current acute or unstable chronic disease other than Postherpetic Neuralgia (PHN)
* Has clinically important medical disorder
* Uses certain types of medications for heart conditions
* Unwilling/unable to discontinue use of medications for treatment of neuropathic pain
* Has a history of hypersensitivity to any medication or soy product
* Has liver or kidney disease
* Has asthma that required treatment within the last year
* Has HIV or hepatitis (other than hepatitis A)
* Has a history of alcohol abuse within the past 2 years
* Has a history of (within last 2 years) or currently abuses prescription or illegal drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Difference (PID) scores (derived from data obtained using the 11 point Likert pain rating scale) | During each Treatment Phase Visit
Various pain related assessment | During each Treatment Phase Visit
Clinical Global Impression of Change (CGIC) and Subject Global Impression of Change (SGIC ) scores | At each Treatment Phase Visit

SECONDARY OUTCOMES:
Incidence, intensity, relationship, and seriousness of treatment-emergent AEs by dose and by treatment group.
Treatment-emergent changes in safety assessments
Evaluation of T-62 plasma concentrations | At various timepoints during the study

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Bradenton Research Center, Bradenton, Florida
  - Anchor Research Center, Naples, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Plains Medical Clinic, Fargo, North Dakota
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Crescent Moon Research, Murrells Inlet, South Carolina
  - Odyssey Research, Spokane, Washington